CLINICAL TRIAL: NCT04576832
Title: Mindfulness Training for U.S. Army Senior Leaders
Brief Title: Mindfulness Training for Senior Leaders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to an enrollment strategy change
Sponsor: University of Miami (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amishi Jha, Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20201075; W911QY-17-C-0101 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Cognitive Change
Keywords: mindfulness training; psychological health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (MT group) (Experimental): Participants will receive 4 weeks of mindfulness training during the first training interval between the first (T1) and second (T2) assessment sessions.
  Interventions: Behavioral: Mindfulness-Based Attention Training (MBAT) web-course
- Group B (Wait-list group) (Active Comparator): Participants will not receive 4 weeks of mindfulness training during the first training interval; they will receive 4 weeks of mindfulness training during the second training interval between the second (T2) and third (T3) assessment sessions.
  Interventions: Behavioral: Mindfulness-Based Attention Training (MBAT) web-course

INTERVENTIONS:
Behavioral: Mindfulness-Based Attention Training (MBAT) web-course — Pre-recorded weekly sessions for 4 weeks. Each session will consist of approximately 2 hours of video content per week and weekly mindfulness exercises. This video will include MBAT program lectures, pre-recorded testimony from military leaders, and teaching materials. The course will also include 15-min daily mindfulness practice drills.

SUMMARY:
The overarching goal of the project is to investigate if a mindfulness-based attention training (MBAT) program contextualized for Military Senior Leaders (SLs) might benefit SLs in three key domains: (1) cognitive abilities, (2) psychological well-being and self-reported physical health, and (3) strategic leadership skills and ability. The MBAT-SL program will be tested by the training cohorts and compared to the wait-list control cohorts who will receive the training after a no-training interval.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are between 18 and 65 years of age.
2. Individuals who are fluent English speakers.
3. Individuals who are active-duty service members
4. Individuals who are willing and able to consent to participate in the study.
5. Individuals who participated in the courses provided by the Army War College (AWC).

Exclusion Criteria:

1. Individuals who have been hospitalized for psychological/mental health issues within the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Change in Sustained attention to response task (SART) score | Baseline (T1) to post-4-week training interval (T2).
  The SART involves pressing a button to frequently presented non-target trials (numbers 1, 2, 4, 5, 6, 7, 8, and 9) and withholding the button press to the infrequent target trials (number 3). The participants can have a total score between 0 and 100% with a higher score indicating better sustained attention.

SECONDARY OUTCOMES:
Change in 5FMQ scores | Baseline (T1) to post-4-week training interval (T2).
  Five-Facet Mindfulness Questionnaire (5FMQ) is used to assess the five major aspects of mindfulness. The present study will use the 15-item short version. The scores range from 15 to 75, with higher scores indicating greater levels of mindfulness in different aspects of one's life.
Change in Decentering score | Baseline (T1) to post-4-week training interval (T2).
  Decentering consists of 11 items measuring various thoughts and experiences, and the tendency to distance from those. The decentering score ranges from 1 to 55, with a higher score indicating a high level of decentering.
Change in PANAS positive affect score | Baseline (T1) to post-4-week training interval (T2).
  Positive and Negative Affect Scale (PANAS) is a widely used self-reported measure of positive and negative affect. The present study will use a short version with a 5-item positive subscale. The score ranges from 5 to 25 with a higher score indicating a higher positive mood.
Change in PANAS negative affect score | Baseline (T1) to post-4-week training interval (T2).
  Positive and Negative Affect Scale (PANAS) is a widely used self-reported measure of positive and negative affect. The present study will use a short version with a 5-item negative subscale. The score ranges from 5 to 25 with a higher score indicating a higher negative mood.
Change in PSS score | Baseline (T1) to post-4-week training interval (T2).
  Perceived Stress Scale (PSS) is a questionnaire measuring the degree to which situations in one's life are viewed as stressful within the past month. The present study will use the 4-item short version, with the total score ranging from 0 to 16, with a higher score indicating a higher level of perceived stress.
Change in PHQ4 scores | Baseline (T1) to post-4-week training interval (T2).
  Patient Health Questionnaire 4 items (PHQ4) is an ultra-brief 4-item measure of depression and anxiety in the general population with the total score ranging from 0 to 12. Higher score indicates higher level of anxiety and depression.

OTHER OUTCOMES:
Change in Leadership Questionnaire | Baseline (T1) to post-4-week training interval (T2).
  Leadership Questionnaire consists of a set of questions that gather information about the self-reported leadership skills and attitudes of Senior Army leaders.
Change in Anger score | Baseline (T1) to post-4-week training interval (T2).
  Dimensions of Anger Reactions (DAR-5) is a self-report measure of anger frequency, intensity, duration, aggression, and impact on social functioning over the past 4 weeks. The scale includes 4 items with a score range of 5-25. Higher scores indicate greater anger levels.
Change in Marital Satisfaction | Baseline (T1) to post-4-week training interval (T2).
  Marital Satisfaction Questionnaire (MSAT) measures one's satisfaction in their current relationship. The scale includes 4 items with a score range of 3-21. Higher scores indicate greater satisfaction with a current relationship.
Applied Mindfulness Practice | Post-4-week training interval 1 (T2) and post-4-week training interval 2 (T3).
  The Applied Mindfulness Process Scale (AMPS) measures one's daily enactment of mindfulness in daily life. Total score ranges from 0 to 60: a higher score indicates a greater application of mindfulness in everyday life.

CONTACTS AND LOCATIONS:
Overall Officials: Amishi Jha, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No